CLINICAL TRIAL: NCT03347201
Title: Thrombin Generation During Cardiopulmonary Bypass With Titrated Versus Conventional Anticoagulation Management.
Acronym: THROMBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-9761
Record Dates: First submitted 2017-10-12; First posted 2017-11-20 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Surgery
Keywords: Cardiopulmonary bypass, Heparin, Protamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Initial heparin bolus before CPB to be calculated using HMS Plus.
  2. Following commencement of CPB further heparin requirements will be determined using the HMS Plus. ACT's will also be checked whilst on CPB and if falls below 480 seconds, additional heparin will also be given.
  3. Following cessation of CPB the dose of protamine required to reverse residual heparin will be calculated using the HMS Plus.
  Interventions: Device: HMS Plus
- Control Group (No Intervention): Patients in the control arm will undergo routine heparin anticoagulation using a weight based initial dose of 400 units/kg, aiming for an ACT of >480 seconds. Further heparin doses (5000 to 10000 units) will be given if the ACT falls below 480 seconds whilst on bypass. At the end of CPB heparin will be reversed with protamine using 1:1 ratio based on the initial dose of heparin given pre-bypass. HMS Plus measures will also be conducted in this group for study purposes, but the results will not be made available to the clinicians.

INTERVENTIONS:
Device: HMS Plus — Subjects randomized to the intervention group will have their dose of Heparin and Protamine calculated by the HMS Plus.
  Arms: Intervention Group

SUMMARY:
In this study, the investigators will be comparing anticoagulation for Cardiopulmonary Bypass (CPB) guided by the Hemostasis Management System (HMS Plus) with the current dosing based on weight and ACT measurements.

The primary objective of this study is to determine whether relative to patients with conventional management, those managed with the HMS Plus have improved thrombin generation after CPB.

The secondary objective is to determine if patients in the HMS Plus group have reduced blood loss in the first 24 hours following surgery compared with patients in the conventional group.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) allows cardiac surgery to be performed on a motionless, bloodless heart while maintaining circulation to the rest of the body. Anticoagulation with heparin prevents the body's clotting system from being activated when blood comes into contact with the walls of the bypass circuit. The amount of heparin given to achieve this effect is determined on a weight-based dosing and monitored with a point-of-care monitor called ACT (activated clotting time). However, there remains a high level of variability in the concentration of heparin in the blood and the ACT is affected by hypothermia and dilution of the blood, both of which commonly occur during CPB for cardiac surgery.

The Hemostasis Management System (HMS Plus) offers an alternative way of dosing and monitoring heparin by aiming to achieve a pre-determined heparin concentration throughout CPB, rather than being determined by the ACT. It also aims to determine the dose of protamine, the drug used to reverse heparin at the end CPB, required based on residual heparin concentration rather than on a 1:1 ratio of the total dose of heparin given which is the common current practice. The benefits of using this system are proposed to be more effective anticoagulation during CPB meaning less of the body's reserves of clotting factors are consumed. This could mean potentially less bleeding and decrease requirement of blood products following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo non-emergent coronary artery bypass grafting, valve repair or replacement (with or without ascending aortic replacement) or a combination of these procedures requiring the use of CPB

Exclusion Criteria:

* Less than 18 years old
* Planned use of deep hypothermic circulatory arrest
* Cases where use of brief circulatory arrest anticipated
* Highly complex cases (LVAD, Heart Transplant, Complex congenital)
* Significant liver dysfunction (liver enzymes > 2-fold higher than upper limit of normal
* Pre-existing coagulopathy (INR >1.5, PTT >45 seconds, fibrinogen < 1.0g/L, platelet count <100x109/L)
* Use of long acting oral anticoagulants
* Patients on heparin infusions pre-operatively
* Major hemoglobinopathies, thalassemia or iron storage diseases
* Previous diagnosis of HIT
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Thrombin Generation | Intra-operative
  The primary outcomes will be thrombin generation potential assessed via peak thrombin and endogenous thrombin potential on CAT thrombograms of plasma samples taken before, during and after cardiopulmonary bypass.

SECONDARY OUTCOMES:
Rotational thromboelastometry (ROTEM) | Intra-operative
  Rotational thromboelastometry will be performed on the ROTEM delta instrument using citrated whole blood.
Activated Clotting Time (ACT) | Intra-operative
  ACTs are performed during surgery
Platelet Function Analysis (PFA) | Intra-operative
  PFA will be performed
Blood loss | Intraoperative day to the 7th postoperative day inclusive
  Amount of blood loss
Blood product transfusion | Intraoperative day to the 7th postoperative day inclusive
  Collection of blood products transfused

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Li H, Bartoszko J, Serrick C, Rao V, Karkouti K. Titrated versus conventional anticoagulation management for thrombin generation in cardiac surgery: a randomized controlled trial. Can J Anaesth. 2022 Sep;69(9):1117-1128. doi: 10.1007/s12630-022-02278-1. Epub 2022 Jul 8. PMID 35799088